CLINICAL TRIAL: NCT01833364
Title: A Pilot Study to Evaluate the Safety and Feasibility of Implanting Autologous Peripheral Nerve Grafts Into the Substantia Nigra of Subjects With Parkinson's Disease Undergoing Deep Brain Stimulation Surgery and Treatment
Brief Title: Autologous Peripheral Nerve Grafts Into the Substantia Nigra of Subjects With PD Undergoing Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig van Horne, MD, PhD (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Craig van Horne, MD, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1021-F6A; 12-1021 (Other: UK CCTS)
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Deep Brain Stimulation; Peripheral Nerve Graft
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantation of Perpherial Nerve Graft (Experimental): Subjects own peripheral nerve tissue that will be used to create the graft for implantation. The autologous peripheral nerve graft will then be implanted unilaterally into the substantia nigra of the subject after the placement of DBS electrodes.
  Interventions: Procedure: Implantation of the Peripheral Nerve Graft

INTERVENTIONS:
Procedure: Implantation of the Peripheral Nerve Graft — The preparatory surgery for harvesting the peripheral nerve graft will take place in the operating room at the time of the Stage I surgery for the DBS procedure. The nerve exposure and preparation will take approximately 15 minutes of operating time in addition to the DBS procedure which typically takes 75-90 minutes.
  The implantation of the nerve graft will take place in the operating room at the end of the second stage surgery for DBS. The graft harvesting and implantation will take approximately 15 minutes in addition to the 4 hours that is needed for the DBS surgery. The subject's peripheral nerve graft will be implanted into the substantia nigra unilaterally. This is a single arm trial to assess safety and feasibility.
  Other Names: Peripheral Nerve Graft

SUMMARY:
By doing this study, the investigators hope to learn provide safety data that can be used to generate a larger phase III clinical trial. If successful, it would promote the development of a new treatment for PD in which patients are able to provide their own tissue as a source of a supportive environment for the injured and dying cells and thereby possibly stopping the progression of the illness or even improve the symptoms of PD.

The purpose of this research is to gather information on the safety and feasibility of nerve graft implantation is. The results of this study will be shared with the University of Kentucky, Center for Clinical and Translational Science (group providing financial support for the study) and other federal agencies, if required.

The overall goal of this research is to develop a novel, regenerative treatment strategy for idiopathic Parkinson's disease (PD) that is safe, cost effective and widely available to patients.

DETAILED DESCRIPTION:
This pilot study is designed to test the safety and feasibility of the implantation of the subject's own peripheral nerve tissue into an area of the brain called the substantia nigra. Only subjects who have elected to undergo DBS surgery will be asked to participate in this research study.

The implantation of the nerve graft will take place in the operating room at the end of the second stage surgery for DBS. Subjects will be asked to donate a piece of their own peripheral nerve tissue that will be used to create the graft for their implantation. The peripheral nerve tissue is obtained from a small incision (approximately 2 inches) above and on the outer-side of one ankle. The initial incision is created during stage I of the DBS procedure and will take place under general anesthesia. The incision will be closed with internal sutures, and a dressing will cover the incision after the procedure.

The nerve will be harvested during stage II of the DBS procedure. This involves opening the same incision using local anesthesia injected around the incision site. Once a small piece (about an inch) of the nerve is removed, the incision will be sutured closed with internal stitches. These stitches will dissolve on their own and will not need to be removed in the office.

Follow-up. Subjects will be followed in our clinic for for DBS follow-up visits and treatment, none of those visits are part of this study.

Prior to coming in for study visits subjects will need to stop taking their PD medications 12 hours before each visit. Subjects will be allowed to restart their normal PD medication during the examination.

Subjects will undergo formal Unified Parkinson's Disease Rating Scale (UPDRS) evaluations at screening and months 1, 3, 6, 9 and 12. In order to visually document potential changes in their Parkinson's Disease symptoms following their DBS surgery, we will be videotaping study related neurological testing sessions.

Subject will also be videotaped at screening, and visits 1, 3, 6, 9, 12.

A neuropsychological exam will be performed at screening and again at month 12.

ELIGIBILITY:
Inclusion Criteria:

* Elected to have DBS Surgery
* Parkinson's Disease for 5 years or more
* Ages 40-75

Exclusion Criteria:

* Have previously undergone PD surgery or any intracranial surgery
* Unwilling to delay taking PD medications during the study
* Unable to follow the directions of the study team
* Unable to attend all study visits
* Have participated in previous clinical studies and received an investigational product within 30 days of screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Nerve Graft Implantation | One year
  All Adverse events will be collected from the time subject signs the consent to the time they complete study visit 12 in order to measure the safety and tolerability of the grafting procedure. Adverse events will be documented and compared to the known and reported adverse events of DBS of STN. In addition, MRI imaging of the graft site within the substantia nigra will be compared to the contralateral, non-grafted site.

SECONDARY OUTCOMES:
Peripheral Nerve Graft Efficacy -- clinical improvement | 1 year
  Post operative data will be collected at study visit 1, 3, 6, 9 and 12 from the time of the second stage surgery.
  * Subjects will undergo UPDRS evaluation at each visit. This will include evaluations with the patients off medication and off stimulation as well as on medication and on stimulation. Comparisons will be evaluated for changes relating to time from implantation as well as between the implanted side vs the non-implanted side.
Peripheral Nerve Graft Efficacy -- Therapy Reduction | 1 year
  This is a composite evaluation targeting changes in medication requirements and DBS stimulation requirements.
  - Changes in medication dosages and stimulation parameters will be recorded at each visit (1,3,6,9,and 12 months post-implantation). Stimulation parameter changes will be evaluated from time of implantation and also compared between the grafted and non-grafted side.
Peripheral Nerve Graft Efficacy -- Quality of Life | 1 year
  Subjects will also have a formal neuropsychological and PDQ-8 examination pre-operatively and at 12 months post implantation. These tests will be used to evaluate psychological profiles and for possible changes in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Craig van Horne, MD, Principal Investigator — University of Kentucky, Department of Neurosurgery
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

REFERENCES:
- [Derived] van Horne CG, Quintero JE, Slevin JT, Anderson-Mooney A, Gurwell JA, Welleford AS, Lamm JR, Wagner RP, Gerhardt GA. Peripheral nerve grafts implanted into the substantia nigra in patients with Parkinson's disease during deep brain stimulation surgery: 1-year follow-up study of safety, feasibility, and clinical outcome. J Neurosurg. 2018 Dec 1;129(6):1550-1561. doi: 10.3171/2017.8.JNS163222. Epub 2018 Feb 18. PMID 29451447
- [Derived] van Horne CG, Quintero JE, Gurwell JA, Wagner RP, Slevin JT, Gerhardt GA. Implantation of autologous peripheral nerve grafts into the substantia nigra of subjects with idiopathic Parkinson's disease treated with bilateral STN DBS: a report of safety and feasibility. J Neurosurg. 2017 Apr;126(4):1140-1147. doi: 10.3171/2016.2.JNS151988. Epub 2016 May 6. PMID 27153166